CLINICAL TRIAL: NCT03278418
Title: Echo-Guided Tricuspid Valve Surgery Vs. Conservative Approach At The Time Of Left- Sided Valve Surgery. A Prospective Randomized Study
Brief Title: Echo-Guided Tricuspid Valve Surgery Vs. Conservative Approach
Acronym: RIGHT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ettore Sansavini Health Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESREFO 32
Record Dates: First submitted 2017-08-31; First posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Tricuspid Valve Insufficiency
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tricuspid Valve Repair (Experimental): Concomitant tricuspid valve repair in patients undergoing left-sided valve surgery
  Interventions: Procedure: Tricuspid Valve Repair; Procedure: Left-sided valve surgery
- left-sided valve surgery (Active Comparator): No concomitant tricuspid valve repair in patients in pts undergoing left-sided valve surgery
  Interventions: Procedure: Left-sided valve surgery

INTERVENTIONS:
Procedure: Tricuspid Valve Repair — It will be performed according to the surgeon preference
  Arms: Tricuspid Valve Repair
Procedure: Left-sided valve surgery — It will be performed according to the surgeon preference

SUMMARY:
Patients elected to undergo any type of left-sided valve surgery (either repair or replacement) with non severe tricuspid regurgitation and tricuspid annular dilation will be screened. Consenting patients fulfilling all inclusion and exclusion criteria will be included in the study and assigned to elective left-sided valve replacement or repair with or without concomitant tricuspid valve repair in a 1:1 fashion, using a blocked randomization scheme balanced within center.

DETAILED DESCRIPTION:
The present study is designed as a prospective, multicentre, multinational, randomized, 2-arm parallel group trial. Participating centres are selected based on previous experience with the surgical technique and standardised echo imaging. Each center is expected to contribute 70 patients over a 12 months enrolment period.

Patients elected to undergo any type of left-sided valve surgery (either repair or replacement) with non severe tricuspid regurgitation and tricuspid annular dilation will be screened. Consenting patients fulfilling all inclusion and exclusion criteria will be included in the study and assigned to elective left-sided valve replacement or repair with or without concomitant tricuspid valve repair in a 1:1 fashion, using a blocked randomization scheme balanced within center.

After discharge patients will be assessed at 1, 12, 24 and 36 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing left-sided valve surgery for left-sided valve disease
* Presence of non-severe TR and tricuspid annular dilation (>40 mm or > 21 mm/m2 BSA) determined by echocardiography
* Age ≥ 18 years
* Capability to sign Informed Consent and Release of Medical Information forms

Exclusion Criteria:

* Preoperative severe TR
* Structural / organic tricuspid valve disease
* Tricuspid annulus ≤40 mm (or ≤ 21 mm/m2 BSA) on preoperative TTE
* Implanted pacemaker or defibrillator, where the leads cross the tricuspid valve from the right atrium into the RV
* Any type of reoperative surgery
* Concomitant cardiac surgery other than atrial fibrillation correction surgery (pulmonary vein isolation, Maze procedure, left atrial appendage closure) or closure of patent foramen ovale or atrial septal defect (for example, concomitant coronary artery bypass graft or aortic surgery)
* Cardiogenic shock at the time of randomization
* ST-elevated myocardial infarction requiring intervention within 7 days prior to randomization
* Evidence of cirrhosis or hepatic synthetic failure
* Severe, irreversible pulmonary hypertension in the judgment of the investigator
* Pregnancy at the time of randomization
* Any concurrent disease with life expectancy < 1 year
* Patient unable or unwilling to provide informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Significant TR (moderate or severe) | 3 years
  To compare in a prospective and randomized way the effect of two different strategies on significant TR (moderate or severe) in patients undergoing surgery for left heart valve disease of any type as assessed by the Core lab evaluation of the echocardiogram. In the echocardiogram images TR by jet area will be grouped as moderate (5-10 cm2) or severe (>10 cm2).

SECONDARY OUTCOMES:
Significant TR (moderate or severe) | 1 and 2 years
  To compare in a prospective and randomized way the effect of two different strategies on significant TR (moderate or severe) in patients undergoing surgery for left heart valve disease of any type as assessed by the Core lab evaluation of the echocardiogram. In the echocardiogram images TR by jet area will be grouped as moderate (5-10 cm2) or severe (>10 cm2).
Mild TR | 1,2 and 3 years
  To compare in a prospective and randomized way the effect of two different strategies on significant TR (moderate or severe) in patients undergoing surgery for left heart valve disease of any type as assessed by the Core lab evaluation of the echocardiogram. In the echocardiogram images TR by jet area will be grouped as non severe (≤10 cm2) or mild (<5 cm2).
Overall TR (mild, moderate, severe) | 1, 2 and 3 years
  To compare in a prospective and randomized way the effect of two different strategies on significant TR (moderate or severe) in patients undergoing surgery for left heart valve disease of any type as assessed by the Core lab evaluation of the echocardiogram. In the echocardiogram images TR by jet area will be grouped as non severe (≤10 cm2; mild <5 cm2, moderate = 5-10 cm2), or severe (>10 cm2).
RV function | 1, 2 and 3 years
  To compare the effect of the 2 strategies for non-severe TR described above on the evaluation of reverse right ventricle (RV) remodelling, assessed as reduction/modification of the end diastolic and end systolic RV diameters.
Pulmonary Artery Pressure (PAP) | 1, 2 and 3 years
  To compare the effect of the 2 strategies for non-severe TR on pulmonary artery pressure (PAP)
Event free survival | 3 years
  Safety evaluation will rely on all AE/SAEs subsequent to spontaneous reporting, or to detection of clinically relevant abnormalities on physical examinations, vital signs, ECG, and laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Maria Salomone, MD, Study Director — Fondazione Ettore Sansavini per la Ricerca Scientifica ONLUS
Locations (4):
- Italy (4):
  - Maria Cecilia Hospital, Cotignola, Ravenna
  - IRCCS Policlinico San Donato, Milan
  - IRCCS Opsedale San Raffaele, Milan
  - Maria Eleonora Hospital, Palermo

IPD SHARING:
Plan to Share IPD: No